CLINICAL TRIAL: NCT07308288
Title: ImmuneNutrition Against Pediatric Respiratory Allergies: Results From the INAPRA Trial
Brief Title: Immune Nutrition in Pediatric Respiratory Allergy
Acronym: INAPRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Full professor, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 104/24
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Asthma Acute; Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study product (Experimental): Intervention
  Interventions: Dietary Supplement: AllergySTOP
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: AllergySTOP — Sodium butyrate FOS (Fructooligosaccharides) Vitamin D3 Heat-inactivated L. rhamnosus GG (LGG) DHA Powder Perilla frutescens Quercetin
  Arms: Study product
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Respiratory allergic diseases, namely asthma and allergic rhinitis (AR), are among the most common chronic pediatric conditions with prevalence continuing to rise over last decades and are leading healthcare costs. Epidemiological trends show high rates in young children, aged under 10 years, significant comorbidity between conditions (asthma and AR), and a rising recognition of lifestyle's role in microbial, epithelial barrier and immune system dysfunction which collectively drive type 2-driven airway inflammation, the hallmark feature of allergic respiratory diseases.

Strategies aiming to reduce allergy outcomes have included dietary interventions during the pediatric age with immunonutrition and postbiotics. Immunonutrition uses specific nutrients to support the immune system, while postbiotics use microbial-derived compounds to modulate microbiome, epithelial barrier and immune function, and they can work together by modulating the gut-immune axis to reduce inflammation and to promote immune tolerance also through epigenetic mechanisms.

Vitamin D, DHA, quercetin, perilla frutescens, fructooligosaccharides and DHA have been indicated as promising food supplements for and effective immunonutrition action against allergy. Similarly, postbiotics-non-viable microbial preparations with demonstrated biological activity-such as heat-inactivated Lactobacillus rhamnosus GG (LGG) and the gut microbiome-derived metabolite butyrate have been shown to strengthen epithelial barrier integrity, modulate cytokine secretion, and promote regulatory immune responses.

Collectively, these findings suggest that targeted nutritional or microbial-derived interventions capable of reinforcing epithelial barrier function and restoring regulatory immune pathways may offer a promising adjunctive strategy for pediatric allergic airway diseases. Despite the expanding mechanistic evidence, clinical trials evaluating multi-component immunomodulatory nutritional interventions in children with asthma or allergic rhinitis remain scarce, and the translational relevance of these mechanistic pathways has not yet been thoroughly tested in controlled pediatric studies.

Based on this rationale, we designed a clinical study to evaluate the clinical and immunological effects of a multi-component supplement containing immunonutritional compounds and postbiotics focusing on symptom control and immunoregulatory biomarkers in PBMCs from children with allergic asthma and AR.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of asthma and/or allergic rhinitis

Exclusion Criteria:

* non-Caucasian ethnicity,
* age <4 or >12 years,
* known hypersensitivity to any of the ingredients of the study product,
* the presence of chronic systemic diseases,
* immunodeficiencies,
* ongoing allergen immunotherapy,
* treatment with immunomodulators,
* systemic corticosteroids, antibiotics, or pre/pro/synbiotics within the four weeks prior to enrollment and during the 6-month study period,
* participation in other studies,
* any condition deemed by the investigators to interfere with study participation or study outcomes.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in respiratory symptom control | after 6 months
  The primary outcome was the change in respiratory symptom control from T0 to T6, assessed using the c-ACT for asthma, and the CARATkids and TNSS for AR.

SECONDARY OUTCOMES:
assessment in PBMCs of IL-4, IL-5, IL-13, IL-10, regulatory T cells (CD4⁺CD25⁺FoxP3⁺), and the expression of tolerogenic dendritic cell-associated markers (Tgfb1, Ifna2, Ptgs2) | at abseline
  at T0, the assessment of immune responses in PBMCs, specifically cytokine secretion profiles (IL-4, IL-5, IL-13, IL-10), the frequency of regulatory T cells (CD4⁺CD25⁺FoxP3⁺), and the expression of tolerogenic dendritic cell-associated markers (Tgfb1, Ifna2, Ptgs2, Csf2)

CONTACTS AND LOCATIONS:
Locations (1):
- Programma Infradipartimentale di Allergologia Pediatrica, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No